CLINICAL TRIAL: NCT00407550
Title: A Randomized Phase II Study of ALIMTA® (Pemetrexed) and GEMZAR® (Gemcitabine) Every 14 Days Versus Pemetrexed and Gemcitabine Every 21 Days in Advanced Non-Small Cell Lung Cancer
Brief Title: Pemetrexed Disodium and Gemcitabine in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000516012; P30CA015083 (NIH); RC0524 (Other: Mayo Clinic Cancer Center & MCCRC); 06-002282 (Other: Mayo Clinic IRB); H3E-US-S061 (Other: Lilly Protocol)
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Results first posted 2012-06-13 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2016-04

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemzar x2 (Experimental): Treat subjects with 2 dosings/cycle of Gemzar x6 cycles.
  Interventions: Drug: gemcitabine HCL; Drug: pemetrexed disodium
- Gemzar x1 (Experimental): Treat subjects with 1 dosing/cycle of Gemzar x9 cycles.
  Interventions: Drug: pemetrexed disodium; Drug: gemcitabine HCL

INTERVENTIONS:
Drug: gemcitabine HCL — 1250 mg/m^2 administered through 250 cc NS (normal saline) IV (intravenous) infusion over 30 minutes at days 1 & 8 of each cycle (21 days) x6 cycles.
  Other Names: GEMZAR
  Arms: Gemzar x2
Drug: pemetrexed disodium — 500 mg/m^2 administered through 100 mL NS IV infusion over 10 minutes at day 1 of each cycle.
  Other Names: ALIMTA
Drug: gemcitabine HCL — 1500 mg/m^2 administered through 250 cc NS IV infusion over 30 minutes at days 1 of each cycle (14 days) x9 cycles.
  Other Names: GEMZAR
  Arms: Gemzar x1

SUMMARY:
RATIONALE: Pemetrexed disodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving pemetrexed disodium together with gemcitabine may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying two different schedules of pemetrexed disodium and gemcitabine to compare how well they work in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare response rates in patients with stage IIIB or IV non-small cell lung cancer treated with two different treatment schedules of pemetrexed disodium and gemcitabine hydrochloride.

Secondary

* Compare time-to-event efficacy variables in patients treated with these regimens.
* Compare progression-free and overall survival of patients treated with these regimens.
* Determine the overall toxicity of these regimens in these patients.

OUTLINE: This is a multicenter, open-label, randomized study. Patients are stratified according to disease stage (IIIB vs IV) and ECOG performance status (0 vs 1). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive pemetrexed disodium IV over 10 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive pemetrexed disodium IV over 10 minutes and gemcitabine hydrochloride IV over 30 minutes on day 1. Treatment repeats every 14 days for up to 9 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 2 years.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IIIB (with controlled pleural effusion) OR stage IV disease
* At least 1 measurable lesion whose longest diameter is ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No medically significant third-space fluid collection (e.g., ascites or pleural effusions) that cannot be controlled by drainage or other procedures
* No documented brain metastases unless all of the following criteria are met:

  * Successful local therapy has been completed
  * At least 2 weeks since prior corticosteroids
  * Brain imaging required for symptomatic patients only (to rule out brain metastases)
* Concurrent enrollment in clinical trial MCCRC-RC0527 required

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 12 weeks
* ECOG performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN
* AST and ALT ≤ 3 times ULN (5 times ULN for liver involvement)
* Creatinine clearance ≥ 45 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to take folic acid, cyanocobalamin (vitamin B12) supplementation, or dexamethasone and corticosteroids
* Able to interrupt intake of aspirin and nonsteroidal anti-inflammatory agents for a total of 5 days
* No severe and/or uncontrolled medical conditions, including any of the following:

  * Hypertension, labile hypertension, or history of poor compliance with antihypertensive medication
  * Angina pectoris
  * Congestive heart failure within the past 3 months, unless ejection fraction > 40%
  * Myocardial infarction within the past 6 months
  * Cardiac arrhythmia
  * Diabetes
  * Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
  * New York Heart Association class III or IV heart disease
  * Clinically significant infection
* No other serious medical condition or illness that would preclude study participation
* No peripheral neuropathy ≥ grade 2
* No other malignancy within the past 5 years except nonmelanomatous skin cancer, carcinoma in situ of the cervix, or low-grade (Gleason score ≤ 6) localized prostate cancer
* No significant weight loss (≥ 10%) within the past 6 weeks
* No investigator site personnel directly affiliated with the study, or immediate family (i.e., spouse, parent, child, or sibling, whether biological or legally adopted)
* No employees of Eli Lilly (i.e., employees, temporary contract workers, or designees responsible for conducting the study)

  * Immediate family of Eli Lilly employees may participate in Eli Lilly-sponsored clinical trials, but are not permitted to participate at an Eli Lilly facility

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 2 weeks since prior corticosteroids
* At least 4 weeks since prior radiation therapy involving > 25% of the bone marrow and recovered
* At least 30 days since prior investigational therapy
* No prior radiation therapy to the whole pelvis
* No prior systemic chemotherapy for advanced non-small cell lung cancer
* No prior pemetrexed disodium and/or gemcitabine hydrochloride
* No prior or concurrent sorafenib tosylate and/or temsirolimus
* No concurrent Hypericum perforatum (St. John's wort)
* No other concurrent antitumor therapy
* No concurrent agents that stimulate thrombopoiesis
* Concurrent palliative radiation therapy allowed
* Concurrent corticosteroids allowed for adrenal insufficiency or severe nausea and vomiting

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2008-01 (Actual); Study Completion 2010-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Molina, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Cancer Center, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 19 patients were enrolled from 9 medical clinics between November 3, 2006 and August 10, 2007.
Period: Overall Study
Arm/Group | Gemzar x2 | Gemzar x1
Started | 10 | 9
Completed | 7 | 5
Not Completed | 3 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Death | 1 | 0
Not completed — Insurance or Other medical condition | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemzar x2 | Gemzar x1 | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Median (Full Range); unit: Years] | 70.5 [60 to 81] | 63 [48 to 74] | 66 [48 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19
Performance Score [Number; unit: Participants] — Classifies patients according to their functional impairment. Scores range from 0 (fully active) to 5 (death).
  Participants
    0 - Fully Active | 4 | 4 | 8
    1 - Ambulatory, restricted strenuous activity | 6 | 5 | 11
Lung Stage [Number; unit: Participants] — From the American Joint Committee on Cancer Staging Criteria for Lung Cancer> N3 - (Regional Lymph Nodes) Metastasis to contralateral mediastinal, contralateral hilar, ipsilateral or contralateral scalene, or supraclavicular lymph nodes(s).> T4 - (Primary Tumor) Tumor of any size that invades any of the following: mediastinum, heart, great vessels, trachea, esophagus, vertebral body, carina; or separate tumor nodules in the same lobe; or tumor with malignant pleural effusion.
  Participants
    IV - Distant Metastasis | 8 | 7 | 15
    IIIB w/pleural effusion - N3 or T4 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Confirmed Responses
Description: Confirmed tumor response (complete and partial) as measured by RECIST(Response Evaluation Criteria In Solid Tumors) criteria on 2 consecutive evaluations at least 6 weeks apart.
  >
  > Confirmed tumor response is at least a 30% decrease in the sum of the longest diameter of target lesions and no new lesions.
Time Frame: Two consecutive evaluations at least 6 weeks apart (up to 2 years)
Measure: Number; unit: participants
Arm/Group | Gemzar x2 | Gemzar x1
Number analyzed (Participants) | 10 | 9
participants | 2 | 0

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the number of months from registration to the date of disease progression or death, with patients who are alive and progression free being censored on the date of their last evaluation.
Time Frame: Time from registration to progression or death (up to 2 years)
Population: One patient in Arm B was deemed a protocol violation and was not include din this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemzar x2 | Gemzar x1
Number analyzed (Participants) | 10 | 8
months | 1.66 [0.69 to 4.3] | 5.04 [1.74 to 5.95]
Statistical Analysis 1: Comparison: Gemzar x2 vs Gemzar x1; Test type: Superiority; p = 0.015, Log Rank

3. Secondary Outcome: Overall Survival
Description: Overall survival time was defined as the number of months from registration to the date of death or last follow-up
Time Frame: Death or last follow-up (up to 2 years)
Population: One patient in Arm B was a major violation and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemzar x2 | Gemzar x1
Number analyzed (Participants) | 10 | 8
months | 5.1 [2.14 to 14.2] | 8.1 [5.5 to 10.1]
Statistical Analysis 1: Comparison: Gemzar x2 vs Gemzar x1; Test type: Superiority; p = 0.56, Log Rank

4. Secondary Outcome: Adverse Event
Description: Number of patients that experienced adverse events (grade 4 or more) as measured by NCI CTCAE (Common Terminology Criteria for Adverse Events) v3.0
Time Frame: Gemzar x2 Arm every 21 days, Gemzar x1 Arm every 14 days (up to 2 years)
Population: All patients that began protocol treatment are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemzar x2 | Gemzar x1
Number analyzed (Participants) | 10 | 9
Participants | 6 | 4

ADVERSE EVENTS:
Arm/Group | Gemzar x2 | Gemzar x1
Serious Adverse Events (participants affected / at risk) | 4/10 | 5/9
Other Adverse Events (participants affected / at risk) | 10/10 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemzar x2 (N=10) | Gemzar x1 (N=9)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Disease Progression (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Blood Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Skin (cellulites) infection (Infections and infestations) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Leukopenia (Investigations) | 2 (3) | 1 (1)
Lymphopenia (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (5) | 3 (3)
Platelet count decreased (Investigations) | 1 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemzar x2 (N=10) | Gemzar x1 (N=9)
Anemia (Blood and lymphatic system disorders) | 8 (29) | 8 (36)
Edema (Cardiac disorders) | 1 (1) | 0 (0)
Vision-Double (Eye disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (9) | 2 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (11) | 7 (20)
Oral cavity Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (4)
Chills (General disorders) | 1 (1) | 0 (0)
Disease Progression (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (10) | 6 (12)
Pain (General disorders) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Lung (pneumonia) infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Forced expiratory volume decreased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Leukopenia (Investigations) | 9 (27) | 8 (23)
Lymphopenia (Investigations) | 1 (7) | 0 (0)
Neutrophil count decreased (Investigations) | 7 (19) | 8 (29)
Platelet count decreased (Investigations) | 7 (12) | 2 (3)
Vital capacity decreased (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Taste (Nervous system disorders) | 1 (1) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes